CLINICAL TRIAL: NCT07039604
Title: Real-World Study of Percutaneous Pulmonary Artery Denervation (PADN) for the Treatment of Pulmonary Arterial Hypertension (PAH)
Brief Title: Real-World Study of PADN for the Treatment of PAH
Status: Recruiting | Type: Observational
Sponsor: Pulnovo Medical (Wuxi) Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: PADN-PMS
Record Dates: First submitted 2025-06-10; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Hypertension; Hypertension, Pulmonary Arterial
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Enhancor™ Radiofrequency Catheter, Pulnovo Medical (Wuxi) CO., Ltd., Wuxi, Jiangsu, China — PADN: Contrast pulmonary artery (PA) angiography will be performed to localize the pulmonary artery bifurcation level and calculate the PA diameter. Once the anatomy deemed acceptable, the radiofrequency ablation catheter will be introduced into ostium of the left PA and the distal bifurcation area of the main PA. The catheter will be manoeuvred within the PA to allow energy delivery in a circumferential manner to ensure that the electrodes are tightly in contact with the endovascular surface. About three ablations at 45-55 # for 120 seconds each will be performed in ostium of the left PA and the distal bifurcation area of the main PA. For non-atrial fibrillation patients, dual antiplatelet therapy for 1 month after PADN is recommended. Patients with atrial fibrillation should continue new oral anticoagulants and patients who underwent metal valve replacement should continued oral warfarin anticoagulation according to guidelines, which could determined by the physician.

SUMMARY:
Real-World Study of PADN for the Treatment of PAH

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with PAH and received PADN procedure since March 2024.
2. No contraindications to procedure.
3. Able to provide informed consent and authorize use of health/research data.
4. Compliant with treatment and follow-up requirements.

Exclusion Criteria:

None specified.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with pulmonary arterial hypertension (PAH) who have undergone PADN procedure.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical worsening | 1 year
  Clinical worsening events defined as any of the following during the study period:
  1. PAH-related rehospitalization.
  2. Addition of PAH-targeted therapies (increased types/dose of PAH-targeted drugs or diuretics).
  3. ≥10% or ≥30-meter reduction in 6-Minute Walk Distance (6MWD) from baseline.
  4. Atrial septostomy.
  5. Need for lung transplantation.
  6. Cardiovascular death.

SECONDARY OUTCOMES:
WHO Functional Class changes from baseline | 6 months, 1, 2, 3, and 5 years
NT-proBNP/BNP levels from baseline | 6 months, 1, 2, 3, and 5 years
6MWD changes from baseline | 6 months, 1, 2, 3, and 5 years
Incidence of pulmonary infections | Through study completion, an average of 5 years
All-cause death | Through study completion, an average of 5 years
Echocardiographic changes from baseline | 6 months, 1, 2, 3, and 5 years
  Right atrial diameter (RAD)
Echocardiographic changes from baseline | 6 months, 1, 2, 3, and 5 years
  Right ventricular end-diastolic diameter (RVDd)
Echocardiographic changes from baseline | 6 months, 1, 2, 3, and 5 years
  Tricuspid annular plane systolic excursion (TAPSE)
Echocardiographic changes from baseline | 6 months, 1, 2, 3, and 5 years
  Left ventricular ejection fraction (LVEF)
Echocardiographic changes from baseline | 6 months, 1, 2, 3, and 5 years
  Left atrial diameter (LAD)
Echocardiographic changes from baseline | 6 months, 1, 2, 3, and 5 years
  Left ventricular end-diastolic diameter (LVDd)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China